CLINICAL TRIAL: NCT07270328
Title: A Pilot Study of Feasibility and Exploratory Study for a Definitive Randomised Controlled Trial of Foot-Ankle Versus Walking Exercises in Patients With Diabetes Mellitus: Effects on Neuropathy, Stress, and Quality of Life
Brief Title: A Pilot Study of the Effectiveness of Foot-Ankle and Walking Exercises in Patients With Diabetes Mellitus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Medical University (Other)
Responsible Party: Principal Investigator, Siti Fadlilah, Principal Investigator, Taipei Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PilotStudyRCT024_Siti Fadlilah
Record Dates: First submitted 2025-11-17; First posted 2025-12-08 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Diabete Mellitus; Diabete Type 2; Diabetic Peripheral Neuropathy; Diabetic Foot; Diabetes; Diabetes (DM); Exercise
Keywords: Diabetic Peripheral Neuropathy; Stress; Quality of life; Fasting blood glucose; Body mass index; Blood pressure; Ankle-brachial index; Diabetes mellitus; Exercise; Waliking exercise; Foot-ankle exercise
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2; Diabetic Foot; Motor Activity | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: Three arms parallel group design with 2 group interventions (foot-ankle exercise and walking exercise) and 1 control group
Who Masked: Outcomes Assessor
Masking Description: Data collectors who assess the outcomes and statistician who analyse the data are blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Foot-ankle exercise group (Experimental): The group received intervention through health education, simulations and leaflets about footankle exercise and practised independently for 12 weeks
  Interventions: Behavioral: Foot-ankle exercise group
- Walking exercise group (Experimental): The group received intervention through health education, and leaflets about walking exercise and practised independently for 12 weeks
  Interventions: Behavioral: Walking exercise group
- Control Group (Active Comparator): The group that received intervention in the form of health education and leaflets about DM in general
  Interventions: Other: Control group

INTERVENTIONS:
Behavioral: Foot-ankle exercise group — Participants in the foot-ankle exercise group received usual care provided by the PHC and an additional intervention consisting of diabetes and foot-ankle exercise education plus a printed leaflet. During the initial session, participants were instructed on the foot-ankle exercise procedures and practiced each movement under supervision to ensure correct technique.
  Following the initial training, participants performed the foot-ankle exercises independently for 12 weeks. One exercise session required approximately 10-15 minutes. To meet the recommended target of moderate physical activity (150 minutes per week), participants were advised to complete 2-3 sessions per day. Participants were instructed to avoid two consecutive days without performing the exercises.
  Participants recorded all home-based foot-ankle exercise sessions on log sheets provided at the first meeting. Intervention monitoring was conducted through regular communication via a moderated group chat.
  Arms: Foot-ankle exercise group
Behavioral: Walking exercise group — Participants in the walking exercise group received usual care provided by the PHC and an additional intervention consisting of diabetes and walking-exercise education plus a printed leaflet. Participants performed walking exercises independently without supervision for 12 weeks.
  Participants were instructed to walk at their usual, comfortable daily pace. The physical activity target was to achieve a moderate level of physical activity totaling 150 minutes per week. To meet this target, participants were advised to complete walking sessions of at least 10 minutes per session, avoid two consecutive days without walking, and ensure a minimum cumulative duration of 150 minutes per week.
  Participants documented all walking-exercise sessions using log sheets provided at the first meeting. Intervention monitoring was conducted through regular communication via a moderated group chat.
  Arms: Walking exercise group
Other: Control group — Usual care and health education Participants in the control group received the usual care provided by the community health center and intervention in the form of health education about DM in general.
  Arms: Control Group

SUMMARY:
This pilot feasibility and exploratory study, conducted to prepare for a definitive Randomized Controlled Trial (RCT), compares a structured foot-ankle exercise program with a walking exercise program in adults with Diabetes Mellitus (DM). The primary aim is to assess feasibility, including recruitment rate, retention, adherence, data completeness, acceptability, and adverse events, to inform procedures for the definitive RCT. The secondary (exploratory) aim is to obtain preliminary estimates of effects on Diabetic Peripheral Neuropathy (DPN), stress, and obstacles to Diabetes-Related Quality of Life (DR-QoL), Fasting Blood Glucose (FBG), Body Mass Index (BMI), blood pressure, and Ankle-Brachial Index (ABI).

Participants were allocated to three parallel arms for 12 weeks:

1. Foot-ankle exercise (education plus printed materials; independent practice 2-3 sessions/day),
2. Walking exercise (education plus printed materials; ≥150 minutes/week, ≥10 minutes/session, avoiding two consecutive non-exercise days), or
3. Active control (education and printed materials).

Outcomes were assessed at baseline (day 0), week 6, and week 12. Analyses focus on feasibility metrics against pre-specified progression criteria and on hypothesis-generating estimates of within- and between-group change in neuropathy, stress, and obstacles to DR-QoL; the study is not powered for definitive efficacy.

Retrospective registration note: This study was registered retrospectively after participant enrolment had begun and data collection had been completed. This retrospective status is disclosed for transparency; exploratory outcome analyses are interpreted accordingly, and adverse events related to exercise were monitored and reported.

DETAILED DESCRIPTION:
Intervention Description Foot-Ankle Exercise Intervention The intervention is adapted from prior research and from exercises developed by the Indonesian Endocrinology Association. Participants receive brief DM and foot-ankle education, a leaflet, and supervised simulation to ensure correct technique. Independent practice is performed 2-3 sessions/day for 12 weeks. Target exercises ≥150 minutes/week.

The structured foot-ankle exercise program consists of 10 seated movements involving toe flexion, heel raises, circular ankle motions, knee extension with toe mobility, synchronized bilateral movements, and functional foot tasks (e.g., manipulating newspaper sheets).

Walking Exercise Intervention The walking program adapts protocols from previous studies. Participants receive DM and walking-exercise education plus a leaflet. They walk independently for ≥150 minutes per week (≥10 minutes/session) while avoiding two consecutive non-exercise days during the 12-week period.

Active Control Participants receive usual DM education (30 minutes) and a leaflet. No structured exercise program is provided.

All groups continue receiving standard public-health services. Weekly monitoring and adverse-event checks are performed.

Content Validity Procedures

A content-validity assessment was conducted to ensure standardization of intervention procedures, educational materials, and measurement protocols (foot sensation, vibration, height, weight, blood pressure, ABI). Six experts (physicians or nurses with ≥5 years of DM-related experience) completed item-level ratings using a 1-4 scale. Content Validity Index (CVI) thresholds:

Item-level (I-CVI) ≥ 0.80 Scale-level (S-CVI) ≥ 0.83 Items below threshold were revised based on expert feedback until satisfactory CVI values were achieved. The CVI results showed I-CVI of >0.90 and S-CVI of 0.96.

Participant Recruitment Recruitment was conducted in partnership with the District Health Office and three Public Health Centers (PHCs) in Yogyakarta operating the Chronic Disease Management Program (PROLANIS). PHCs identified potentially eligible adults with DM and supported initial contact. Interested individuals received standardized information regarding study procedures, risks/benefits, confidentiality, and voluntary participation. Those willing attended a screening and informed-consent session. After consent, participants were enrolled and added to the communication group.

Participants received travel reimbursement of IDR 25,000 per data-collection visit. Recruitment materials were approved by the Institutional Review Board (IRB). Participation was voluntary and did not affect access to routine services.

Sample Size A total of 108 participants (36 per group) were enrolled, accounting for an estimated 20% attrition rate. Sample size was selected for feasibility assessment and to provide preliminary, hypothesis-generating estimates for DPN, stress, and DR-QoL outcomes; it was not used to determine the sample size of the subsequent definitive RCT.

Actual Completion Numbers Week 6: control n=35, foot-ankle n=35, walking n=33 Week 12: control n=32, foot-ankle n=34, walking n=34 Per-protocol: control n=31, foot-ankle n=33, walking n=31

Randomization and Allocation Concealment Randomization was performed by independent personnel not involved in recruitment or data collection. A computer-generated sequence with random permuted blocks (sizes 3, 6, and 9) was used with a 1:1:1 allocation ratio.

Assignments were placed in sequentially numbered, sealed, opaque envelopes stored securely and inaccessible to outcome assessors..

Intervention Delivery Control group The active control group was given health education on the topic of DM for 30 minutes and then given a leaflet.

Foot-ankle exercise group

Participants were given health education on DM and foot-ankle exercise after the allocation procedure, followed by simulation and practice lasts 60 minutes. Participants were also given leaflets. Afterward, participants practiced independently without supervision for 12 weeks. Foot-ankle exercise consists of 10 movements. When doing foot-ankle exercises, participants sit comfortably without leaning, and the soles of their feet touch the floor and barefoot. These movements are:

A 1. Lift the soles while heels touch the floor. 2. Flex toes downward (clawing motion). 3. Repeat 10 times. B

1. Lift the soles while heels touch the floor.
2. Lower soles and raise heels while toes touch the floor.
3. Repeat 10 times. C

<!-- -->

1. Lift the soles while heels touch the floor.
2. Perform inward-to-outward circular motions.
3. Repeat 10 times. D

1. Lift both heels while toes touch the floor. 2. Perform inward-to-outward circular motions. 3. Repeat 10 times. E

1. Lift and extend the right knee; left leg remains in original position.
2. Move toes forward and backward.
3. Repeat 10 times; repeat on left leg. F

<!-- -->

1. Lift and extend the right knee.
2. Move toes toward the face.
3. Repeat 10 times; repeat on left leg. G

<!-- -->

1. Lift and extend both knees.
2. Move toes toward the face simultaneously.
3. Repeat 10 times. H

<!-- -->

1. Lift and extend both knees.
2. Move both legs forward.
3. Repeat 10 times. I

<!-- -->

1. Lift and extend the right knee; left leg remains in place.
2. "Write" numbers 1-10 using the right foot.
3. Repeat with the left foot. J

1. Place a sheet of newspaper under both feet. 2. Crumple into a ball using both feet. 3. Open it back into a sheet. 4. Tear into two parts using both feet. 5. Tear one part into small pieces and gather onto the other sheet. 6. Crumple into a ball again. 7. Dispose of the newspaper ball in the trash.

Walking exercise group Participants were given health education for 30 minutes, on DM and walking exercises and leaflet after the allocation procedure. Participants practiced walking exercises independently for 12 weeks.

Health education for all groups is delivered by a certified DM educator. To minimize contamination, group education is conducted on separate days. All participants are added to a moderated WhatsApp group for communication, scheduling, and reminders..

Interventionist dan Outcome Investigators

Interventions are delivered by a health professional with:

- a master's degree in nursing,

* ≥5 years of clinical/educator experience, and
* certification as a DM educator. Each site includes ≥1 outcome investigator who is a registered health worker.

Monitor for Adverse Events Potential adverse events included fatigue, muscle soreness, pain, and dizziness. Participants self-recorded events and reported them during weekly telephone monitoring. If excessive or concerning adverse events were identified, the intervention was stopped and appropriate care provided.

ELIGIBILITY:
Inclusion Criteria:

* People with type 2 diabetes
* Aged 20-70 years
* Diagnosed with DM for at least 1 year
* Can walk without assistance
* Able to communicate well
* Can read and write
* Willing to be a respondent

Exclusion Criteria:

* Has a history of leg amputation
* Have a diagnosis of heart failure, kidney failure, pulmonary TB, stroke
* Patients with a history or under-treatment of mental disorders
* DM patients with foot ulcers
* DM patients with fractures or difficulty using the lower extremities

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2024-07-05 (Actual); Primary Completion 2024-09-29 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Feasibility: Recruitment Rate | From July 5, 2024 (first participant enrollment) to September 29, 2024 (final primary outcome data collection), over an actual period of approximately 12 weeks.
  Participants enrolled per month per site and overall; eligibility and consent proportions
Feasibility: Retention Rate | From July 5, 2024 (Baseline assessment) to September 29, 2024 (Week 12 follow-up), over an actual period of approximately 12 weeks.
  Proportion of enrolled participants who complete follow-up assessments at Week 6 and Week 12.
Feasibility: Adherence to Assigned Intervention | From July 5, 2024 (Week 0, baseline) to September 29, 2024 (Week 12 assessment), covering an actual intervention period of approximately 12 weeks.
  Percentage of prescribed sessions achieved (foot-ankle and walking exercise) with ≥150 min/week and "no two consecutive non-exercise days"; proportion meeting adherence threshold (≥70%) across ≥12 weeks
Feasibility: Data Completeness | From July 5, 2024 (Baseline) to September 29, 2024 (Week 12 follow-up), covering the period in which data completeness at Week 6 and Week 12 was assessed (12 weeks).
  Proportion of participants with complete outcome data at Week 6 and Week 12 (per arm and overall).
Feasibility: Safety (Adverse Events) | From July 5, 2024 (start of intervention at Week 0) to September 29, 2024 (Week 12 follow-up), covering an actual 12-week period of adverse event monitoring.
  Exercise-related adverse events/serious adverse events (number and percentage)
Feasibility: Acceptability of the Intervention (Open-Ended Participant Feedback) | From July 5, 2024 (start of intervention) to September 29, 2024 (Week 12), when acceptability feedback was collected, covering an actual period of approximately 12 weeks.
  Open-ended questions elicit participants' messages/impressions, barriers, and difficulties during the intervention. Responses will be analysed with rapid thematic analysis using a pre-defined codebook; two independent coders will code all transcripts/notes, discrepancies resolved by discussion

SECONDARY OUTCOMES:
Diabetic Peripeheral Neuropathy (DPN) | From July 5, 2024 (Baseline) to September 29, 2024 (Week 12), during which DPN was assessed at Baseline, Week 6, and Week 12; covering an actual 12-week period.
  DPN measured by Michigan Neuropathy Scale Instrument (MNSI). MNSI consist of MNSI-A (questionnaire) and MNSI-B (physical examination). Foot sensation was measured by Semmes Weinstein Monofilament 10g. Participants were given a stimulus for 1.5-2 seconds at 10 points on both legs. The locations are heel, dorsal surface (between the bases of 1st-2nd toes), toes (1st, 3rd and 5th), metatarsal heads (1st, 3rd, 5th), and midfoot (medial and lateral). The results range from 0-10. Foot vibration measurement using Tunning Fork 128Hz. The vibrating TF were placed on each leg in 4 locations (medial, malleolus, great toe, fifth toe). Participants were asked to feel the vibrations and signal by raising their hands if they were no longer felt. The observer recorded the time from when the participant feels the initial until it disappears. The results consist of whether the participant felt the vibration or not (0-4) and the length of time participants can feel the vibration (in seconds).
Stress | From July 5, 2024 (Baseline) to September 29, 2024 (Week 12), during which stress was assessed at Baseline, Week 6, and Week 12 over an actual 12-week period.
  Stress was measured using the Indonesian version of the Problem Areas in Diabetes (PAID) questionnaire. This study used PAID Bahasa Indonesia, which we have previously tested for validity and reliability. PAID Bahasa Indonesia has 20 items and three factors, with a loading factor of 0.349-0.779 for each item. The results of exploratory factor analysis (EFA) and confirmatory factor analysis (CFA) show valid and reliable results. Cronbach's alpha for all items is 0.858, inter-class correlation 0.938, RMSEA=0.058, and SRMR=0.062. PAID Bahasa Indonesia consist of five answer choices using a Likert scale (0-4). The answer choice scores used were 'not a problem' (0), 'minor problem' (1), 'moderate problem' (2), 'somewhat serious problem' (3), and 'serious problem' (4). The total score ranged 0-100, with a higher score indicating greater stress.
Obstacles to Diabetes Related Quality of Life (DR-QoL) | From July 5, 2024 (Baseline) to September 29, 2024 (Week 12), during which DR-QoL (DOQ-30) was assessed at Baseline, Week 6, and Week 12 over an actual 12-week period.
  Obstacles to DR-QoL measured using the Indonesian version of the Diabetes Obstacles Questionnaire Short Version (DOQ-30) which we have previously tested for validity and reliability. Factors in the DOQ-30 are relationships with medical professionals, support from friends and family, knowledge of the disease, lifestyle changes, exercising, self-monitoring, uncertainty about a consultation, medication, and insulin use. EFA and CFA analysis showed valid and reliable results; Cronbach's alpha for all items was 0.930, and individual factors ranged from 0.730 to 0.848. The test-retest results were excellent (with interclass correlation coefficients of 0.910 to 0.973). The CFA test obtained RMSEA=0.057 and SRMR=0.067, indicating a good model fit. The DOQ-30 contains nine domains and 30 items rated on a 0-4 Likert scale ("never" to "always"), with scores standardized from 0 (no obstacles) to 1 (worst possible obstacles).
Fasting Blood Glucose (FBG) | From July 5, 2024 (Baseline) to September 29, 2024 (Week 12), during which fasting blood glucose was measured at Baseline, Week 6, and Week 12 over an actual 12-week period.
  FBG were measured using venous blood after the respondent fasted for at least 8 hours. Blood analysis is carried out in the laboratory using the hexokinase enzymatic method. The researchers did not carry out this analysis, but they collaborated with the Independent Clinical Laboratory. All participants were measured according to standard operating procedures as a guide. The measurement results are documented in the observation sheet. The process of taking venous blood is carried out by nursing staff with the criteria of having a competency certificate and working for a minimum of 3 years.
Blood Pressure | From July 5, 2024 (Baseline) to September 29, 2024 (Week 12), during which blood pressure was measured at Baseline, Week 6, and Week 12 over an actual 12-week period.
  Blood pressure was measured using a digital tensimeter, The Omron M3 Intellisense (Omron Healthcare Co Ltd), validated in previous research. Participants were asked to rest for at least 5 minutes before the measurement. Measurements were taken on the left arm in a sitting or supine position. Blood pressure consists of Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP) in mmHg units. Then, the mean atrial pressure (MAP) will be calculated using the formula, MAP = DBP + 1/3(SBP - DBP) or MAP = DBP + 1/3(pulse pressure/PP) All participants were measured according to standard operating procedures as a guide. The measurement results are documented in the observation sheet.
Body Mass Index (BMI) | From July 5, 2024 (Baseline) to September 29, 2024 (Week 12), during which BMI was measured at Baseline, Week 6, and Week 12 over an actual 12-week period.
  Participants were asked to stand up straight and remove footwear when their height and weight were checked. Body weight was measured using digital scales, and height using height-measuring devices. BMI is calculated using the formula body weight (kg) divided by height2 (m2). All participants were measured according to standard operating procedures as a guide. The measurement results are documented in the observation sheet
Ankle-Brachial Index (ABI) | From July 5, 2024 (Baseline) to September 29, 2024 (Week 12), during which ABI was measured at Baseline, Week 6, and Week 12 over an actual 12-week period.
  ABI measurements carried out using continuous-wave Doppler ultrasound. Participants were asked to rest for at least 5 minutes, and measurements were taken in the supine position. Blood pressure was measured twice each at four locations: right arm, left arm, right leg and left leg. Arm blood pressure was measured by Doppler ultrasound in the humeral artery, while leg blood pressure was placed in the tibial artery. The cuff is inflated 20-30 mmHg and deflated slowly. The first sound heard is systolic blood pressure. The average blood pressure results from the two measurements at each location will be calculated to obtain the average blood pressure in the right arm, left arm, right leg and left leg. ABI calculated using the ankle SBP/brachial SBP formula. The results of these calculations produce the right and left ABI.

CONTACTS AND LOCATIONS:
Overall Officials: Siti Fadlilah, Principal Investigator — Taipei Medical University
Locations (3):
- Indonesia (3):
  - Puskesmas Ngaglik 1, Sleman, Special Region of Yogyakarta
  - Puskesmas Ngemplak 1, Sleman, Special Region of Yogyakarta
  - Puskesmas Ngemplak 2, Sleman, Special Region of Yogyakarta

IPD SHARING:
Plan to Share IPD: Yes
Particular data will be shared: Individual participant data that underlie the results reported in this article after identification (text, tables, figures, and appendices).
Supporting Information: Study Protocol
Time Frame: Beginning 9 months and ending 60 months following article publication.
Access Criteria: Investigators whose proposed use of the data has been approved by an independent review committee ("learned intermediary") identified for this purpose, for example, for a meta-analysis or other study.

REFERENCES:
- [Background] Henderson AD, Johnson AW, Rasmussen LG, Peine WP, Symons SH, Scoresby KA, Ridge ST, Bruening DA. Early-Stage Diabetic Neuropathy Reduces Foot Strength and Intrinsic but Not Extrinsic Foot Muscle Size. J Diabetes Res. 2020 Mar 12;2020:9536362. doi: 10.1155/2020/9536362. eCollection 2020. PMID 32258170
- [Result] Zhu X, Zhao L, Chen J, Lin C, Lv F, Hu S, Cai X, Zhang L, Ji L. The Effect of Physical Activity on Glycemic Variability in Patients With Diabetes: A Systematic Review and Meta-Analysis of Randomized Controlled Trials. Front Endocrinol (Lausanne). 2021 Nov 17;12:767152. doi: 10.3389/fendo.2021.767152. eCollection 2021. PMID 34867812
- [Result] Zheng ZJ, Rosamond WD, Chambless LE, Nieto FJ, Barnes RW, Hutchinson RG, Tyroler HA, Heiss G; ARIC Investigators. Lower extremity arterial disease assessed by ankle-brachial index in a middle-aged population of African Americans and whites: the Atherosclerosis Risk in Communities (ARIC) Study. Am J Prev Med. 2005 Dec;29(5 Suppl 1):42-9. doi: 10.1016/j.amepre.2005.07.019. PMID 16389125
- [Result] Yuenyongchaiwat K, Pipatsitipong D, Sangprasert P. Increasing walking steps daily can reduce blood pressure and diabetes in overweight participants. Diabetol Int. 2017 Aug 7;9(1):75-79. doi: 10.1007/s13340-017-0333-z. eCollection 2018 Feb. PMID 30603352
- [Result] Young MJ, Breddy JL, Veves A, Boulton AJ. The prediction of diabetic neuropathic foot ulceration using vibration perception thresholds. A prospective study. Diabetes Care. 1994 Jun;17(6):557-60. doi: 10.2337/diacare.17.6.557. PMID 8082524
- [Result] Win MMTM, Fukai K, Nyunt HH, Linn KZ. Hand and foot exercises for diabetic peripheral neuropathy: A randomized controlled trial. Nurs Health Sci. 2020 Jun;22(2):416-426. doi: 10.1111/nhs.12676. Epub 2019 Dec 26. PMID 31876991
- [Result] Whelton SP, Chin A, Xin X, He J. Effect of aerobic exercise on blood pressure: a meta-analysis of randomized, controlled trials. Ann Intern Med. 2002 Apr 2;136(7):493-503. doi: 10.7326/0003-4819-136-7-200204020-00006. PMID 11926784
- [Result] Wang Y, Mou Q, Zhao D, Xu Y, Hu D, Ma H, Liu J, Guo X, Li J. Predictive value of ankle-brachial index and blood glucose on the outcomes of six-year all-cause mortality and cardiovascular mortality in a Chinese population of type 2 diabetes patients. Int Angiol. 2012 Dec;31(6):586-94. PMID 23222938
- [Result] Umpierre D, Ribeiro PA, Kramer CK, Leitao CB, Zucatti AT, Azevedo MJ, Gross JL, Ribeiro JP, Schaan BD. Physical activity advice only or structured exercise training and association with HbA1c levels in type 2 diabetes: a systematic review and meta-analysis. JAMA. 2011 May 4;305(17):1790-9. doi: 10.1001/jama.2011.576. PMID 21540423
- [Result] Tan LS. The clinical use of the 10g monofilament and its limitations: a review. Diabetes Res Clin Pract. 2010 Oct;90(1):1-7. doi: 10.1016/j.diabres.2010.06.021. Epub 2010 Jul 22. PMID 20655123
- [Result] Takahara M, Fujiwara Y, Sakamoto F, Katakami N, Matsuoka TA, Kaneto H, Shimomura I. Assessment of vibratory sensation with a tuning fork at different sites in Japanese patients with diabetes mellitus. J Diabetes Investig. 2014 Feb 12;5(1):90-3. doi: 10.1111/jdi.12126. Epub 2013 Aug 28. PMID 24843743
- [Result] Sartor CD, Hasue RH, Cacciari LP, Butugan MK, Watari R, Passaro AC, Giacomozzi C, Sacco IC. Effects of strengthening, stretching and functional training on foot function in patients with diabetic neuropathy: results of a randomized controlled trial. BMC Musculoskelet Disord. 2014 Apr 27;15:137. doi: 10.1186/1471-2474-15-137. PMID 24767584
- [Result] Saeedi P, Petersohn I, Salpea P, Malanda B, Karuranga S, Unwin N, Colagiuri S, Guariguata L, Motala AA, Ogurtsova K, Shaw JE, Bright D, Williams R; IDF Diabetes Atlas Committee. Global and regional diabetes prevalence estimates for 2019 and projections for 2030 and 2045: Results from the International Diabetes Federation Diabetes Atlas, 9th edition. Diabetes Res Clin Pract. 2019 Nov;157:107843. doi: 10.1016/j.diabres.2019.107843. Epub 2019 Sep 10. PMID 31518657
- [Result] Rias YA, Kurniawan AL, Chang CW, Gordon CJ, Tsai HT. Synergistic Effects of Regular Walking and Alkaline Electrolyzed Water on Decreasing Inflammation and Oxidative Stress, and Increasing Quality of Life in Individuals with Type 2 Diabetes: A Community Based Randomized Controlled Trial. Antioxidants (Basel). 2020 Oct 1;9(10):946. doi: 10.3390/antiox9100946. PMID 33019646
- [Result] Qiu S, Cai X, Schumann U, Velders M, Sun Z, Steinacker JM. Impact of walking on glycemic control and other cardiovascular risk factors in type 2 diabetes: a meta-analysis. PLoS One. 2014 Oct 17;9(10):e109767. doi: 10.1371/journal.pone.0109767. eCollection 2014. PMID 25329391
- [Result] Polonsky WH, Anderson BJ, Lohrer PA, Welch G, Jacobson AM, Aponte JE, Schwartz CE. Assessment of diabetes-related distress. Diabetes Care. 1995 Jun;18(6):754-60. doi: 10.2337/diacare.18.6.754. PMID 7555499
- [Result] Pilv L, Vermeire E, Ratsep A, Moreau A, Nikolic D, Petek D, Yaman H, Oona M, Kalda R. Development and validation of the short version of the diabetes obstacles questionnaire (DOQ-30) in six European countries. Eur J Gen Pract. 2016;22(1):16-22. doi: 10.3109/13814788.2015.1093619. Epub 2015 Nov 18. PMID 26578192
- [Result] Oluchi SE, Manaf RA, Ismail S, Kadir Shahar H, Mahmud A, Udeani TK. Health Related Quality of Life Measurements for Diabetes: A Systematic Review. Int J Environ Res Public Health. 2021 Sep 1;18(17):9245. doi: 10.3390/ijerph18179245. PMID 34501838
- [Result] Monteiro RL, Ferreira JSSP, Silva EQ, Cruvinel-Junior RH, Verissimo JL, Bus SA, Sacco ICN. Foot-ankle therapeutic exercise program can improve gait speed in people with diabetic neuropathy: a randomized controlled trial. Sci Rep. 2022 May 9;12(1):7561. doi: 10.1038/s41598-022-11745-0. PMID 35534614
- [Result] Linderman GC, Lu J, Lu Y, Sun X, Xu W, Nasir K, Schulz W, Jiang L, Krumholz HM. Association of Body Mass Index With Blood Pressure Among 1.7 Million Chinese Adults. JAMA Netw Open. 2018 Aug 3;1(4):e181271. doi: 10.1001/jamanetworkopen.2018.1271. PMID 30646115
- [Result] Lin X, Xu Y, Pan X, Xu J, Ding Y, Sun X, Song X, Ren Y, Shan PF. Global, regional, and national burden and trend of diabetes in 195 countries and territories: an analysis from 1990 to 2025. Sci Rep. 2020 Sep 8;10(1):14790. doi: 10.1038/s41598-020-71908-9. PMID 32901098
- [Result] Lee S, Kim H, Choi S, Park Y, Kim Y, Cho B. Clinical usefulness of the two-site Semmes-Weinstein monofilament test for detecting diabetic peripheral neuropathy. J Korean Med Sci. 2003 Feb;18(1):103-7. doi: 10.3346/jkms.2003.18.1.103. PMID 12589096
- [Result] Kirwan JP, Solomon TP, Wojta DM, Staten MA, Holloszy JO. Effects of 7 days of exercise training on insulin sensitivity and responsiveness in type 2 diabetes mellitus. Am J Physiol Endocrinol Metab. 2009 Jul;297(1):E151-6. doi: 10.1152/ajpendo.00210.2009. Epub 2009 Apr 21. PMID 19383872
- [Result] Islam FMA, Islam MA, Hosen MA, Lambert EA, Maddison R, Lambert GW, Thompson BR. Associations of physical activity levels, and attitudes towards physical activity with blood pressure among adults with high blood pressure in Bangladesh. PLoS One. 2023 Feb 3;18(2):e0280879. doi: 10.1371/journal.pone.0280879. eCollection 2023. PMID 36735692
- [Result] Inzucchi SE, Bergenstal RM, Buse JB, Diamant M, Ferrannini E, Nauck M, Peters AL, Tsapas A, Wender R, Matthews DR. Management of hyperglycemia in type 2 diabetes, 2015: a patient-centered approach: update to a position statement of the American Diabetes Association and the European Association for the Study of Diabetes. Diabetes Care. 2015 Jan;38(1):140-9. doi: 10.2337/dc14-2441. No abstract available. PMID 25538310
- [Result] Ingrosso DMF, Primavera M, Samvelyan S, Tagi VM, Chiarelli F. Stress and Diabetes Mellitus: Pathogenetic Mechanisms and Clinical Outcome. Horm Res Paediatr. 2023;96(1):34-43. doi: 10.1159/000522431. Epub 2022 Feb 4. PMID 35124671
- [Result] Hyun S, Forbang NI, Allison MA, Denenberg JO, Criqui MH, Ix JH. Ankle-brachial index, toe-brachial index, and cardiovascular mortality in persons with and without diabetes mellitus. J Vasc Surg. 2014 Aug;60(2):390-5. doi: 10.1016/j.jvs.2014.02.008. Epub 2014 Mar 21. PMID 24657294
- [Result] Guglani R, Shenoy S, Sandhu JS. Effect of progressive pedometer based walking intervention on quality of life and general well being among patients with type 2 diabetes. J Diabetes Metab Disord. 2014 Nov 29;13(1):110. doi: 10.1186/s40200-014-0110-5. eCollection 2014. PMID 25493265
- [Result] Francia P, Anichini R, De Bellis A, Seghieri G, Lazzeri R, Paternostro F, Gulisano M. Diabetic foot prevention: the role of exercise therapy in the treatment of limited joint mobility, muscle weakness and reduced gait speed. Ital J Anat Embryol. 2015;120(1):21-32. PMID 26738255
- [Result] Ferreira JSSP, Sacco ICN, Siqueira AA, Almeida MHM, Sartor CD. Rehabilitation technology for self-care: Customised foot and ankle exercise software for people with diabetes. PLoS One. 2019 Jun 20;14(6):e0218560. doi: 10.1371/journal.pone.0218560. eCollection 2019. PMID 31220155
- [Result] Faizah R, Efendi F, Suprajitno S. The effects of foot exercise with audiovisual and group support foot exercises to diabetes mellitus patients. J Diabetes Metab Disord. 2021 Feb 22;20(1):377-382. doi: 10.1007/s40200-021-00756-9. eCollection 2021 Jun. PMID 34178845
- [Result] Dube S, Hulke SM, Wakode SL, Khadanga S, Thakare AE, Bharshankar RN, Pakhare A. Effectiveness of Semmes Weinstein 10 gm monofilament in diabetic peripheral neuropathy taking nerve conduction and autonomic function study as reference tests. J Family Med Prim Care. 2022 Oct;11(10):6204-6208. doi: 10.4103/jfmpc.jfmpc_195_22. Epub 2022 Oct 31. PMID 36618173
- [Result] de la Vega R, Jimenez-Castuera R, Leyton-Roman M. Impact of Weekly Physical Activity on Stress Response: An Experimental Study. Front Psychol. 2021 Jan 12;11:608217. doi: 10.3389/fpsyg.2020.608217. eCollection 2020. PMID 33510685
- [Result] Craig AB, Strauss MB, Daniller A, Miller SS. Foot sensation testing in the patient with diabetes: introduction of the quick & easy assessment tool. Wounds. 2014 Aug;26(8):221-31. PMID 25860638
- [Result] Ankle Brachial Index Collaboration; Fowkes FG, Murray GD, Butcher I, Heald CL, Lee RJ, Chambless LE, Folsom AR, Hirsch AT, Dramaix M, deBacker G, Wautrecht JC, Kornitzer M, Newman AB, Cushman M, Sutton-Tyrrell K, Fowkes FG, Lee AJ, Price JF, d'Agostino RB, Murabito JM, Norman PE, Jamrozik K, Curb JD, Masaki KH, Rodriguez BL, Dekker JM, Bouter LM, Heine RJ, Nijpels G, Stehouwer CD, Ferrucci L, McDermott MM, Stoffers HE, Hooi JD, Knottnerus JA, Ogren M, Hedblad B, Witteman JC, Breteler MM, Hunink MG, Hofman A, Criqui MH, Langer RD, Fronek A, Hiatt WR, Hamman R, Resnick HE, Guralnik J, McDermott MM. Ankle brachial index combined with Framingham Risk Score to predict cardiovascular events and mortality: a meta-analysis. JAMA. 2008 Jul 9;300(2):197-208. doi: 10.1001/jama.300.2.197. PMID 18612117
- [Result] Colberg SR, Sigal RJ, Yardley JE, Riddell MC, Dunstan DW, Dempsey PC, Horton ES, Castorino K, Tate DF. Physical Activity/Exercise and Diabetes: A Position Statement of the American Diabetes Association. Diabetes Care. 2016 Nov;39(11):2065-2079. doi: 10.2337/dc16-1728. No abstract available. PMID 27926890
- [Result] Cerrahoglu L, Kosan U, Sirin TC, Ulusoy A. Range of Motion and Plantar Pressure Evaluation for the Effects of Self-Care Foot Exercises on Diabetic Patients with and Without Neuropathy. J Am Podiatr Med Assoc. 2016 May;106(3):189-200. doi: 10.7547/14-095. PMID 27269974
- [Result] Bull FC, Al-Ansari SS, Biddle S, Borodulin K, Buman MP, Cardon G, Carty C, Chaput JP, Chastin S, Chou R, Dempsey PC, DiPietro L, Ekelund U, Firth J, Friedenreich CM, Garcia L, Gichu M, Jago R, Katzmarzyk PT, Lambert E, Leitzmann M, Milton K, Ortega FB, Ranasinghe C, Stamatakis E, Tiedemann A, Troiano RP, van der Ploeg HP, Wari V, Willumsen JF. World Health Organization 2020 guidelines on physical activity and sedentary behaviour. Br J Sports Med. 2020 Dec;54(24):1451-1462. doi: 10.1136/bjsports-2020-102955. PMID 33239350
- [Result] Brown SJ, Handsaker JC, Bowling FL, Boulton AJ, Reeves ND. Diabetic peripheral neuropathy compromises balance during daily activities. Diabetes Care. 2015 Jun;38(6):1116-22. doi: 10.2337/dc14-1982. Epub 2015 Mar 12. PMID 25765355
- [Result] Boulton AJ, Vinik AI, Arezzo JC, Bril V, Feldman EL, Freeman R, Malik RA, Maser RE, Sosenko JM, Ziegler D; American Diabetes Association. Diabetic neuropathies: a statement by the American Diabetes Association. Diabetes Care. 2005 Apr;28(4):956-62. doi: 10.2337/diacare.28.4.956. No abstract available. PMID 15793206
- [Result] Belli T, Ribeiro LF, Ackermann MA, Baldissera V, Gobatto CA, Galdino da Silva R. Effects of 12-week overground walking training at ventilatory threshold velocity in type 2 diabetic women. Diabetes Res Clin Pract. 2011 Sep;93(3):337-43. doi: 10.1016/j.diabres.2011.05.007. Epub 2011 Jun 1. PMID 21636159
- [Result] Battista F, Ermolao A, van Baak MA, Beaulieu K, Blundell JE, Busetto L, Carraca EV, Encantado J, Dicker D, Farpour-Lambert N, Pramono A, Bellicha A, Oppert JM. Effect of exercise on cardiometabolic health of adults with overweight or obesity: Focus on blood pressure, insulin resistance, and intrahepatic fat-A systematic review and meta-analysis. Obes Rev. 2021 Jul;22 Suppl 4(Suppl 4):e13269. doi: 10.1111/obr.13269. Epub 2021 May 6. PMID 33960110
- [Result] Aylin K, Arzu D, Sabri S, Handan TE, Ridvan A. The effect of combined resistance and home-based walking exercise in type 2 diabetes patients. Int J Diabetes Dev Ctries. 2009 Oct;29(4):159-65. doi: 10.4103/0973-3930.57347. PMID 20336198
- [Result] Aschalew AY, Yitayal M, Minyihun A. Health-related quality of life and associated factors among patients with diabetes mellitus at the University of Gondar referral hospital. Health Qual Life Outcomes. 2020 Mar 10;18(1):62. doi: 10.1186/s12955-020-01311-5. PMID 32156282
- [Result] Amin N, Doupis J. Diabetic foot disease: From the evaluation of the "foot at risk" to the novel diabetic ulcer treatment modalities. World J Diabetes. 2016 Apr 10;7(7):153-64. doi: 10.4239/wjd.v7.i7.153. PMID 27076876
- [Result] American Diabetes Association. 2. Classification and Diagnosis of Diabetes: Standards of Medical Care in Diabetes-2021. Diabetes Care. 2021 Jan;44(Suppl 1):S15-S33. doi: 10.2337/dc21-S002. PMID 33298413
- [Result] American Diabetes Association. Standards of medical care in diabetes-2015 abridged for primary care providers. Clin Diabetes. 2015 Apr;33(2):97-111. doi: 10.2337/diaclin.33.2.97. No abstract available. PMID 25897193
- [Result] Aloke C, Egwu CO, Aja PM, Obasi NA, Chukwu J, Akumadu BO, Ogbu PN, Achilonu I. Current Advances in the Management of Diabetes Mellitus. Biomedicines. 2022 Sep 29;10(10):2436. doi: 10.3390/biomedicines10102436. PMID 36289697
- [Result] Adu MD, Malabu UH, Malau-Aduli AEO, Malau-Aduli BS. Enablers and barriers to effective diabetes self-management: A multi-national investigation. PLoS One. 2019 Jun 5;14(6):e0217771. doi: 10.1371/journal.pone.0217771. eCollection 2019. PMID 31166971
- [Result] Aboyans V, Criqui MH, Abraham P, Allison MA, Creager MA, Diehm C, Fowkes FG, Hiatt WR, Jonsson B, Lacroix P, Marin B, McDermott MM, Norgren L, Pande RL, Preux PM, Stoffers HE, Treat-Jacobson D; American Heart Association Council on Peripheral Vascular Disease; Council on Epidemiology and Prevention; Council on Clinical Cardiology; Council on Cardiovascular Nursing; Council on Cardiovascular Radiology and Intervention, and Council on Cardiovascular Surgery and Anesthesia. Measurement and interpretation of the ankle-brachial index: a scientific statement from the American Heart Association. Circulation. 2012 Dec 11;126(24):2890-909. doi: 10.1161/CIR.0b013e318276fbcb. Epub 2012 Nov 16. No abstract available. PMID 23159553
- [Result] Barone Gibbs B, Dobrosielski DA, Althouse AD, Stewart KJ. The effect of exercise training on ankle-brachial index in type 2 diabetes. Atherosclerosis. 2013 Sep;230(1):125-30. doi: 10.1016/j.atherosclerosis.2013.07.002. Epub 2013 Jul 14. PMID 23958264
- [Result] Alqahtani KM, Bhangoo M, Vaida F, Denenberg JO, Allison MA, Criqui MH. Predictors of Change in the Ankle Brachial Index with Exercise. Eur J Vasc Endovasc Surg. 2018 Mar;55(3):399-404. doi: 10.1016/j.ejvs.2017.12.004. Epub 2018 Jan 20. PMID 29371037
- [Result] Alves-Cabratosa L, Comas-Cufi M, Ponjoan A, Garcia-Gil M, Marti-Lluch R, Blanch J, Elosua-Bayes M, Parramon D, Camos L, Guzman L, Ramos R. Levels of ankle-brachial index and the risk of diabetes mellitus complications. BMJ Open Diabetes Res Care. 2020 Mar;8(1):e000977. doi: 10.1136/bmjdrc-2019-000977. PMID 32144131
- [Result] Asfaw MS, Dagne WK. Physical activity can improve diabetes patients' glucose control; A systematic review and meta-analysis. Heliyon. 2022 Dec 13;8(12):e12267. doi: 10.1016/j.heliyon.2022.e12267. eCollection 2022 Dec. PMID 36578408
- [Result] Asmar R, Khabouth J, Topouchian J, El Feghali R, Mattar J. Validation of three automatic devices for self-measurement of blood pressure according to the International Protocol: The Omron M3 Intellisense (HEM-7051-E), the Omron M2 Compact (HEM 7102-E), and the Omron R3-I Plus (HEM 6022-E). Blood Press Monit. 2010 Feb;15(1):49-54. doi: 10.1097/MBP.0b013e3283354b11. PMID 20032779
- [Result] Birke JA, Patout CA Jr, Foto JG. Factors associated with ulceration and amputation in the neuropathic foot. J Orthop Sports Phys Ther. 2000 Feb;30(2):91-7. doi: 10.2519/jospt.2000.30.2.91. PMID 10693087
- [Result] Bonora E, Trombetta M, Dauriz M, Travia D, Cacciatori V, Brangani C, Negri C, Perrone F, Pichiri I, Stoico V, Zoppini G, Rinaldi E, Da Prato G, Boselli ML, Santi L, Moschetta F, Zardini M, Bonadonna RC. Chronic complications in patients with newly diagnosed type 2 diabetes: prevalence and related metabolic and clinical features: the Verona Newly Diagnosed Type 2 Diabetes Study (VNDS) 9. BMJ Open Diabetes Res Care. 2020 Aug;8(1):e001549. doi: 10.1136/bmjdrc-2020-001549. PMID 32819978
- [Result] Boulton AJ, Vileikyte L, Ragnarson-Tennvall G, Apelqvist J. The global burden of diabetic foot disease. Lancet. 2005 Nov 12;366(9498):1719-24. doi: 10.1016/S0140-6736(05)67698-2. PMID 16291066
- [Result] Bus SA, Lavery LA, Monteiro-Soares M, Rasmussen A, Raspovic A, Sacco ICN, van Netten JJ; International Working Group on the Diabetic Foot. Guidelines on the prevention of foot ulcers in persons with diabetes (IWGDF 2019 update). Diabetes Metab Res Rev. 2020 Mar;36 Suppl 1:e3269. doi: 10.1002/dmrr.3269. PMID 32176451
- [Result] Cai H, Li G, Zhang P, Xu D, Chen L. Effect of exercise on the quality of life in type 2 diabetes mellitus: a systematic review. Qual Life Res. 2017 Mar;26(3):515-530. doi: 10.1007/s11136-016-1481-5. Epub 2016 Dec 18. PMID 27990609
- [Result] Childs E, de Wit H. Regular exercise is associated with emotional resilience to acute stress in healthy adults. Front Physiol. 2014 May 1;5:161. doi: 10.3389/fphys.2014.00161. eCollection 2014. PMID 24822048
- [Result] Cho NH, Shaw JE, Karuranga S, Huang Y, da Rocha Fernandes JD, Ohlrogge AW, Malanda B. IDF Diabetes Atlas: Global estimates of diabetes prevalence for 2017 and projections for 2045. Diabetes Res Clin Pract. 2018 Apr;138:271-281. doi: 10.1016/j.diabres.2018.02.023. Epub 2018 Feb 26. PMID 29496507
- [Result] Crawford F, Inkster M, Kleijnen J, Fahey T. Predicting foot ulcers in patients with diabetes: a systematic review and meta-analysis. QJM. 2007 Feb;100(2):65-86. doi: 10.1093/qjmed/hcl140. PMID 17277315
- [Result] Cruvinel-Junior RH, Ferreira JSSP, Verissimo JL, Monteiro RL, Suda EY, Silva EQ, Sacco ICN. Could an Internet-Based Foot-Ankle Therapeutic Exercise Program Modify Clinical Outcomes and Gait Biomechanics in People with Diabetic Neuropathy? A Clinical Proof-of-Concept Study. Sensors (Basel). 2022 Dec 7;22(24):9582. doi: 10.3390/s22249582. PMID 36559949
- [Result] de Boer IH, Bangalore S, Benetos A, Davis AM, Michos ED, Muntner P, Rossing P, Zoungas S, Bakris G. Diabetes and Hypertension: A Position Statement by the American Diabetes Association. Diabetes Care. 2017 Sep;40(9):1273-1284. doi: 10.2337/dci17-0026. No abstract available. PMID 28830958
- [Result] Defay R, Delcourt C, Ranvier M, Lacroux A, Papoz L. Relationships between physical activity, obesity and diabetes mellitus in a French elderly population: the POLA study. Pathologies Oculaires liees a l' Age. Int J Obes Relat Metab Disord. 2001 Apr;25(4):512-8. doi: 10.1038/sj.ijo.0801570. PMID 11319655
- [Result] Dong XL, Guan F, Xu SJ, Zhu LX, Zhang PP, Cheng AB, Liu TJ. Influence of blood glucose level on the prognosis of patients with diabetes mellitus complicated with ischemic stroke. J Res Med Sci. 2018 Jan 29;23:10. doi: 10.4103/1735-1995.223951. eCollection 2018. PMID 29456567
- [Result] Ferrannini E, Cushman WC. Diabetes and hypertension: the bad companions. Lancet. 2012 Aug 11;380(9841):601-10. doi: 10.1016/S0140-6736(12)60987-8. PMID 22883509
- [Result] Gram B, Christensen R, Christiansen C, Gram J. Effects of nordic walking and exercise in type 2 diabetes mellitus: a randomized controlled trial. Clin J Sport Med. 2010 Sep;20(5):355-61. doi: 10.1227/NEU.0b013e3181e56e0a. PMID 20818193
- [Result] Gray N, Picone G, Sloan F, Yashkin A. Relation between BMI and diabetes mellitus and its complications among US older adults. South Med J. 2015 Jan;108(1):29-36. doi: 10.14423/SMJ.0000000000000214. PMID 25580754
- [Result] Hoogendoorn SW, Rutten GEHM, Hart HE, de Wolf C, Vos RC. A simple to implement and low-cost supervised walking programme in highly motivated individuals with or at risk for type 2 diabetes: An observational study with a pre-post design. Prev Med Rep. 2018 Nov 7;13:30-36. doi: 10.1016/j.pmedr.2018.11.003. eCollection 2019 Mar. PMID 30510891
- [Result] Kanade RV, van Deursen RW, Harding K, Price P. Walking performance in people with diabetic neuropathy: benefits and threats. Diabetologia. 2006 Aug;49(8):1747-54. doi: 10.1007/s00125-006-0309-1. Epub 2006 Jun 7. PMID 16758177
- [Result] Kanchanasamut W, Pensri P. Effects of weight-bearing exercise on a mini-trampoline on foot mobility, plantar pressure and sensation of diabetic neuropathic feet; a preliminary study. Diabet Foot Ankle. 2017 Feb 20;8(1):1287239. doi: 10.1080/2000625X.2017.1287239. eCollection 2017. PMID 28326159
- [Result] Karstoft K, Clark MA, Jakobsen I, Muller IA, Pedersen BK, Solomon TP, Ried-Larsen M. The effects of 2 weeks of interval vs continuous walking training on glycaemic control and whole-body oxidative stress in individuals with type 2 diabetes: a controlled, randomised, crossover trial. Diabetologia. 2017 Mar;60(3):508-517. doi: 10.1007/s00125-016-4170-6. Epub 2016 Dec 9. PMID 27942800
- [Result] Kelley GA, Kelley KS. Progressive resistance exercise and resting blood pressure : A meta-analysis of randomized controlled trials. Hypertension. 2000 Mar;35(3):838-43. doi: 10.1161/01.hyp.35.3.838. PMID 10720604
- [Result] Kirwan JP, Sacks J, Nieuwoudt S. The essential role of exercise in the management of type 2 diabetes. Cleve Clin J Med. 2017 Jul;84(7 Suppl 1):S15-S21. doi: 10.3949/ccjm.84.s1.03. PMID 28708479
- [Result] Lu B, Hu J, Wen J, Zhang Z, Zhou L, Li Y, Hu R. Determination of peripheral neuropathy prevalence and associated factors in Chinese subjects with diabetes and pre-diabetes - ShangHai Diabetic neuRopathy Epidemiology and Molecular Genetics Study (SH-DREAMS). PLoS One. 2013 Apr 16;8(4):e61053. doi: 10.1371/journal.pone.0061053. Print 2013. PMID 23613782
- [Result] Rac-Albu M, Iliuta L, Guberna SM, Sinescu C. The role of ankle-brachial index for predicting peripheral arterial disease. Maedica (Bucur). 2014 Sep;9(3):295-302. PMID 25705296
- [Result] Moher D, Hopewell S, Schulz KF, Montori V, Gotzsche PC, Devereaux PJ, Elbourne D, Egger M, Altman DG. CONSORT 2010 explanation and elaboration: updated guidelines for reporting parallel group randomised trials. BMJ. 2010 Mar 23;340:c869. doi: 10.1136/bmj.c869. No abstract available. PMID 20332511
- [Result] Park S, Kim J, Lee J. Effects of Exercise Intervention on Adults With Both Hypertension and Type 2 Diabetes Mellitus: A Systematic Review and Meta-analysis. J Cardiovasc Nurs. 2021 Jan/Feb;36(1):23-33. doi: 10.1097/JCN.0000000000000651. PMID 32011348
- [Result] Schaper NC, van Netten JJ, Apelqvist J, Bus SA, Hinchliffe RJ, Lipsky BA; IWGDF Editorial Board. Practical Guidelines on the prevention and management of diabetic foot disease (IWGDF 2019 update). Diabetes Metab Res Rev. 2020 Mar;36 Suppl 1:e3266. doi: 10.1002/dmrr.3266. PMID 32176447
- [Result] Shah SZA, Karam JA, Zeb A, Ullah R, Shah A, Haq IU, Ali I, Darain H, Chen H. Movement is Improvement: The Therapeutic Effects of Exercise and General Physical Activity on Glycemic Control in Patients with Type 2 Diabetes Mellitus: A Systematic Review and Meta-Analysis of Randomized Controlled Trials. Diabetes Ther. 2021 Mar;12(3):707-732. doi: 10.1007/s13300-021-01005-1. Epub 2021 Feb 5. PMID 33547579
- [Result] Diabetes Canada Clinical Practice Guidelines Expert Committee; Sigal RJ, Armstrong MJ, Bacon SL, Boule NG, Dasgupta K, Kenny GP, Riddell MC. Physical Activity and Diabetes. Can J Diabetes. 2018 Apr;42 Suppl 1:S54-S63. doi: 10.1016/j.jcjd.2017.10.008. No abstract available. PMID 29650112
- [Result] Soleimani Tapehsari B, Alizadeh M, Khamseh ME, Seifouri S, Nojomi M. Physical Activity and Quality of Life in People with Type 2 Diabetes Mellitus: A Randomized Controlled Trial. Int J Prev Med. 2020 Jan 24;11:9. doi: 10.4103/ijpvm.IJPVM_202_18. eCollection 2020. PMID 32089809
- [Result] Suryani M, Samekto W, Heri-Nugroho, Susanto H, Dwiantoro L. Effect of foot-ankle flexibility and resistance exercise in the secondary prevention of plantar foot diabetic ulcer. J Diabetes Complications. 2021 Sep;35(9):107968. doi: 10.1016/j.jdiacomp.2021.107968. Epub 2021 May 28. PMID 34187716
- [Result] Tesfaye S, Boulton AJ, Dyck PJ, Freeman R, Horowitz M, Kempler P, Lauria G, Malik RA, Spallone V, Vinik A, Bernardi L, Valensi P; Toronto Diabetic Neuropathy Expert Group. Diabetic neuropathies: update on definitions, diagnostic criteria, estimation of severity, and treatments. Diabetes Care. 2010 Oct;33(10):2285-93. doi: 10.2337/dc10-1303. PMID 20876709
- [Result] Weinstein AR, Sesso HD, Lee IM, Cook NR, Manson JE, Buring JE, Gaziano JM. Relationship of physical activity vs body mass index with type 2 diabetes in women. JAMA. 2004 Sep 8;292(10):1188-94. doi: 10.1001/jama.292.10.1188. PMID 15353531
- [Result] Welch GW, Jacobson AM, Polonsky WH. The Problem Areas in Diabetes Scale. An evaluation of its clinical utility. Diabetes Care. 1997 May;20(5):760-6. doi: 10.2337/diacare.20.5.760. PMID 9135939
- [Result] Yang MC, Huang YY, Hsieh SH, Sun JH, Wang CC, Lin CH. Ankle-Brachial Index Is Independently Associated With Cardiovascular Outcomes and Foot Ulcers in Asian Patients With Type 2 Diabetes Mellitus. Front Endocrinol (Lausanne). 2021 Nov 18;12:752995. doi: 10.3389/fendo.2021.752995. eCollection 2021. PMID 34867797
- [Result] Herman WH, Pop-Busui R, Braffett BH, Martin CL, Cleary PA, Albers JW, Feldman EL; DCCT/EDIC Research Group. Use of the Michigan Neuropathy Screening Instrument as a measure of distal symmetrical peripheral neuropathy in Type 1 diabetes: results from the Diabetes Control and Complications Trial/Epidemiology of Diabetes Interventions and Complications. Diabet Med. 2012 Jul;29(7):937-44. doi: 10.1111/j.1464-5491.2012.03644.x. PMID 22417277
- See also: International Diabetes Federation, I. (2021). IDF Diabetes Atlas 10th edition. Available IPD/Information: — http://www.diabetesatlas.org